CLINICAL TRIAL: NCT05598814
Title: Optimisation of Treatment in Patients with CRSwNP. an RCT of Mepolizumab and Surgical Treatment with FESS and Mepolizumab Versus Only Mepolizumab Over a 6- and 12-month Follow-up
Brief Title: Mepolizumab to CRSwNP Through 12 Months - Randomised to FESS and Non-FESS Within the First 2 Weeks
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vibeke Backer (Other)
Responsible Party: Sponsor-Investigator, Vibeke Backer, Professor, Pulmonologist, MD, DMSc (PI), Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-ENT-FESS-nonFESS
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-11

CONDITIONS: Chronic Rhinosinusitis with Nasal Polyps; Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: The study is a randomized clinical trial with two arms. Arm 1: Biologic treatment with Mepolizumab every month combined with Arm 2: Only biologic treatment with Mepolizumab every month combined with Functional Endoscopic Sinus Surgery (FESS) 2 weeks after the first injection of Mepolizumab.
Who Masked: Outcomes Assessor
Masking Description: The Nasal Polyp Score (NPS) evaluation will be performed by a third surgeon (blinded evaluation) who will not know the results of the screening visit and FESS/non-FESS randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group - FESS (Experimental): Biologic treatment with Mepolizumab and functional endoscopic sinus surgery (FESS).
  Interventions: Biological: Mepolizumab Injection; Procedure: Functional Endoscopic Sinus Surgery (FESS).
- Control group - No-FESS (Active Comparator): Biologic treatment with Mepolizumab
  Interventions: Biological: Mepolizumab Injection

INTERVENTIONS:
Biological: Mepolizumab Injection — All patients in both the intervention group and the control group will be treated with Mepolizumab injections every month.
Procedure: Functional Endoscopic Sinus Surgery (FESS). — The Functional Endoscopic Sinus Surgery will be performed 2 weeks after the first injection of Mepolizumab in the intervention group.
  Arms: Intervention group - FESS

SUMMARY:
This clinical trial will compare treatment in patients with chronic rhinosinusitis with nasal polyps (CRSwNP) and asthma. The patients will be randomized to treatment with the biologic drug, Mepolizumab, or the biologic drug Mepolizumab combined with Functional Endoscopic Sinus Surgery (FESS).

The aim of this study is to evaluate the effect of combined treatment with biologic treatment and surgery vs. biologic treatment only.

The hypothesis is that surgical removal of polyps and inflamed tissue from the nasal sinuses will increase the effect of the biologic treatment, leading to a lower disease burden after 6 months of treatment, compared with biologic drugs only. Furthermore, combined biologics and surgery will keep a lower disease burden and better general health after 12 months of treatment than biologics alone.

Inclusion criteria:

* Patients ≥ 18 years old at the time of signed informed consent (no upper limit)
* Patients who are referred to the outpatient clinic for the following reasons:

  * Doctor's diagnosis of CRS
* NPS ≥ 2+2 out of a score of 8 (max)
* Severity measured as an SNOT22 score > 35
* One FESS in general anaesthesia performed prior to inclusion (no time limitations)
* No course of systemic steroids within the last 3 months, whereas a daily low dose is allowed
* Possible doctor's diagnosis of asthma
* Type 2 inflammation

Exclusion criteria:

* Patients who, because of language barriers, are not able to understand written information and, thus, are not able to answer questionnaires
* Patients who currently receive biologics for any other disease
* Patients who have previously or currently received biologics for CRS or asthma
* Patients who are not able to give informed consent (i.e., patients who are permanently incapable)
* Patients who meet ≥1 of the following:

  * Malignant lung disease
  * Cardiac disease of clinical importance
  * Current pregnancy and breastfeeding, as well as planning to be pregnant in the near future
  * Unwillingness to have FESS performed
* Patients needing FESS or systemic steroids (OCS) during the study period will be excluded after an unscheduled visit (last observation carried forward (LOCF))
* Patients who are not eligible because of the investigator's judgement

The effect of the treatment will be evaluated with objective procedures and questionnaires related to CRSwNP and asthma after 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old at the time of signed informed consent (no upper limit)
* Patients who are referred to the outpatient clinic for the following reasons:

  * Doctor's diagnosis of CRS
* NPS ≥ 2+2 out of a score of 8 (max)
* Severity measured as an SNOT22 score > 35
* One FESS surgery in general anaesthesia performed prior to inclusion (no time limitations)
* No course of systemic steroids within the last 3 months, whereas a daily low dose is allowed
* Possible doctor's diagnosis of asthma
* Type 2 inflammation

Exclusion Criteria:

* Patients who, because of language barriers, are not able to understand written information and, thus, are not able to answer questionnaires
* Patients who currently receive biologics for any other disease
* Patients who have previously or currently received biologics for CRS or asthma
* Patients who are not able to give informed consent (i.e., patients who are permanently incapable)
* Patients who meet ≥1 of the following:

  * Malignant lung disease
  * Cardiac disease of clinical importance
  * Current pregnancy and breastfeeding, as well as planning to be pregnant in the near future
  * Unwillingness to have FESS performed
* Patients needing FESS or systemic steroids (OCS) during the study period will be excluded after an unscheduled visit (last observation carried forward (LOCF))
* Patients who are not eligible because of the investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in The Sino-Nasal Outcome Test 22 (SNOTT22) score | 6 months
  The success rate indicated by a significant change in health-related quality of life related to nasal symptoms measured with the questionnaire SNOT22. The outcomes to be evaluated are the differences in success rates between the two treatment arms Minimum score = 0 and maximum score = 110 with high scores indicating a large rhinosinusitis-related health burden.

SECONDARY OUTCOMES:
Change in Vo2max/kg(Cardiopulmonary exercise test ) | 6 and 12 motnhs folow-up
  Highest oxygen consumption measured on a stationary ergometer bike divided by body weight. MCID: 1 ml/min/kg
Change in Daily step count | 6 and 12 months follow up
  Measured as an average daily step count over 7 days using a smartphone
Change in Activity level(questionnaire) | 6 and 12 months follow up
  Patient's self-reported amount of exercise, measured using a questionnaire (customised AQUA)
Change in Nasal Polyp Score (NPS) | 3 and 6 months follow up
  The NPS scale ranges from 0 (no polyp) to 4 (large polyps) for each nostril. The total score ranging from 0-8.
Change in Forced Expired Volume in the first second (FEV1) | 6 and 12 months follow up
  Change in Forced Expired Volume in the first second (FEV1). The value is corrected for age, sex, height and weight.
Change in forced vital capacity (FVC) | 3, 6, and 12 months follow up
  The value is corrected for age, sex, height and weight.
Change in Asthma Control Questionnaire (ACQ) score | 3, 6, and 12 months follow up
  Change in ACQ-score. Minimum score = 0 and maximum score = 6 with high scores indicating a large asthma-related health burden.
Change in ratio between FEV1/FVC | 3, 6, and 12 months follow up
  FEV1 divided by FVC. A ratio <0.70 is considered as obstructive.
Change in nitric oxide in exhaled air | 6 and 12 months follow up
  Change in nitric oxide in exhaled air examined with Exhaled Nitric Oxide Test (FeNO). A value between 0-25 is normal. A value >25 indicates inflammation in the airways.
Change in middle ear pressure | 12 months
  Change in middle ear pressure examined with a tympanometry. A =normal, B= flat curve, fluid or perfusion, C1= negative pressure down to -150 dPa, C2 = negative pressure below -150 dPA.
Change in olfactory function | 6 and 12 months follow up
  Change in olfactory function measured with Sniffin' Sticks Identification Test 16.
  Minimum score = 0. Maximum score = 16. A score between 0-8 indicates anosmia, a score between 8-11 indicates hyposmia, and a score >11 indicates normosmia.
Change in Functional Outcomes of Sleep Questionnaire (FOSQ) score | 3, 6, and 12 months follow up
  FOSQ-10 consists of 10 questions rated on a scale of 1 to 4 (1=extreme difficulty and 4=no difficulty).
Change in Epworth Sleepiness score (ESS) | 3, 6, and 12 months follow up
  ESS consists of 8 questions rated on a scale of 0 to 3 (3=extreme difficulty and 0=no difficulty)
Change in AHI/ODI | 6, and 12 months follow up
  Measurement of objective sleep parameters (Apnea hypopnea index and Oxygen desaturation index)
Change in Blood Eosinophilic cell count | 3, 6, and 12 months follow up.
  Blood Eosinophilic cell count from full blood cell count (109/mL).
Change in Polyp Eosinophilic cell count | 6 and 12 months follow up.
  Tissue eosinophilia, classified into four categories: none (0), mild (<10 hpf), moderate (10-100 hpf), and severe (>100 hpf).
Change in Small airway dysfunction | 6 and 12 months follow up.
  Measured by the average flow from the point at which 25 percent of the FVC has been exhaled to the point at which 75 percent of the FVC has been exhaled(MFEF75/25) and Impulse oscillometry: Difference in R5Hz and R20Hz , AX and X5Hz.
Change in Bronchial hyperresponsiveness | 6 and 12 months follow up
  Assessed through methacholine and mannitol challenge tests. Methacholine inhalation ranged from 0 to 1440 µg, with a positive test defined as a ≥20% decrease in FEV1 (PD20). Mannitol inhalation ranged from 0 to 635 mg, with a positive test defined as a ≥15% decrease in FEV1 (PD15)
Change in eosinophilic cell count in sputum | 6 and 12 months follow up
  Sputum induced through the inhalation of hypertonic saline at increasing concentrations (3%, 4%, and 5%). Percentual amount of Eosinophilic cells.
Change in NasalNO | 6 and 12 months follow up
  A value greater then 255-300 is considered normal, whereas values less than 77 nl/min is abnormal.
Change in visual analogue scale (VAS) | 3, 6, and 12 months follow up
  Change in VAS related to nasal symptoms. Minimum score = 0 and maximum score = 10. High score indicates worse nasal symptoms
Change in visual analogue scale (VAS) | 3, 6, and 12 months follow up
  Change in VAS related to asthma symptoms. Minimum score = 0 and maximum score = 100. High score indicates worse Asthma symptoms
Change in visual analogue scale (VAS) | 3, 6 and 12 months follow-up
  Change in VAS related to Smell. Minimum score = 0 and maximum score = 100. High score indicates worse Hyposmia Symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke B Backer, Professor, Study Chair — Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Rigshospitalet
Locations (1):
- Rigshospitalet, Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Copenhagen, Denmark